CLINICAL TRIAL: NCT02972424
Title: PTH(1-34) and Pelvic Fracture Healing - a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-330
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Results first posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Osteoporotic Fractures
Keywords: pelvic fracture; healing; teriparatide
MeSH Terms: conditions — Osteoporotic Fractures; Hip Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teriparatide Prefilled Syringe (Experimental): TPTD is supplied as a sterile, colorless, clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable delivery device (pen) for subcutaneous injection. Each prefilled delivery device is filled with 2.7 mL to deliver 2.4 mL. Each mL contains 250 mcg teriparatide (corrected for acetate, chloride, and water content), 0.41 mg glacial acetic acid, 0.1 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3 mg Metacresol, and Water for Injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4.
  Interventions: Drug: Teriparatide Prefilled Syringe
- Placebo (Placebo Comparator): Placebo is supplied as a sterile, colorless, clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable delivery device (pen) for subcutaneous injection. Each prefilled delivery device is filled with 2.7 mL to deliver 2.4 mL. Each mL contains 0.41 mg glacial acetic acid, 0.1 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3 mg Metacresol, and Water for Injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide Prefilled Syringe — TPTD 20 mcg
  Other Names: Forteo
  Arms: Teriparatide Prefilled Syringe
Drug: Placebo — Matching placebo as a prefilled syringe with all inactive ingredients
  Other Names: Placebo prefilled syringe
  Arms: Placebo

SUMMARY:
In the proposed trial the investigators will recruit women and men >65 years of age with acute osteoporosis-related pelvic fractures and address 3 specific aims over 3 months of treatment in a placebo controlled double blind study to determine if standard care and teriparatide 20 mcg/day versus placebo for pelvic fractures:

1. Results in earlier evidence of cortical bridging on routine radiographs followed by confirmatory Focus CT, a novel method to reduce radiation exposure from CT scans (primary outcome).
2. Leads to a faster reduction in pain as assessed by both the Numeric Rating Scale and a reduction in the use of narcotics (secondary outcome).
3. Leads more rapidly to improved functional outcome using a short physical performance battery to assess lower extremity function (secondary outcome).

DETAILED DESCRIPTION:
The incidence rate of pelvic fractures increases dramatically with age, from 5.4 and 3.8 per 10,000 person-years in women and men aged 65 to 69 years to 93.5 and 44.5 per 10,000 person-years in women and men aged 90 years and older, respectively. Pelvic fractures are accompanied by severe pain, chronic immobility and loss of function and independence in the elderly. Pelvic fractures consume substantial healthcare resources, and based on administrative claims data, they are one of the most costly osteoporosis related fractures. Un-healed fractures, occurring in one-third of pelvic fracture patients at 3 months, can cause continued pain and impact mobility. With aging of the population, and expected concomitant increase in the incidence of pelvic fractures, there is a pressing need to find effective treatments that will accelerate healing. Fracture of the pubic ramus is most relevant and practical for randomized double-blinded placebo controlled study as this fracture is accompanied by severe pain and immobility in elderly, is associated with delayed fracture healing, and is almost always treated non-operatively. The current standard of care for pelvic fractures includes pain management, patient mobilization, and the prevention of complications associated with comorbid conditions. The investigators hypothesize that development of a successful adjunctive therapy to accelerate fracture healing would lead to improved care and reduce both direct and indirect costs from pelvic fractures. In the proposed trial the investigators will recruit women and men >65 years of age with acute osteoporosis-related pelvic fractures and address 3 specific aims over 3 months of treatment in a placebo controlled double blind study to determine if standard care and teriparatide 20 mcg/day versus placebo for pelvic fractures:

1. Results in earlier evidence of cortical bridging on routine radiographs followed by confirmatory Focus CT, a novel method to reduce radiation exposure from CT scans (primary outcome).
2. Leads to a faster reduction in pain as assessed by both the Numeric Rating Scale and a reduction in the use of narcotics (secondary outcome).
3. Leads more rapidly to improved functional outcome using a short physical performance battery to assess lower extremity function (secondary outcome).

The investigators will extend this study with 9 months of open label TPTD to determine if any potential differences between the placebo and TPTD groups during the 3 months of treatment are evident and persist over time, even in patients who use TPTD after the three month placebo controlled intervention. If TPTD can improve fracture healing, this study will have an impact on the treatment of persons with pelvic fracture who are not surgical candidates and often face severe pain, chronic immobility, and loss of function in the elderly. A positive finding of accelerated healing of pelvic fractures would also encourage study of TPTD for treatment of other osteoporotic fractures.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women and men >65 years of age with acute pelvic fractures, occurring with minimal trauma, presenting to Helen Hayes Hospital, Hospital for Special Surgery, or New York Hospital (Cornell Medical). Patients that have either one or multiple pelvic fractures or sacral and pelvic fractures will be included in the study. Subjects must start treatment within one month of hip fracture.

Exclusion Criteria:

1. Persons unable to complete the NRS and other surveys based on their mini-mental status score (≤18; consistent with moderate and severe cognitive impairment)
2. Previously (prior to fracture) non-ambulatory subjects
3. Exclusion criteria related to contraindication or intolerance to TPTD:

   1. Hypersensitivity to TPTD
   2. Patients with increased risk of osteosarcoma: Paget's disease, history of radiation exposure
   3. Patients with active hypercalcemia
   4. Current hyperparathyroidism and other metabolic bone disease including osteogenesis imperfecta
   5. History of multiple renal calculi or renal calculus within the last 2 years
   6. Normal alkaline phosphatase levels will not be used as an entrance criterion because most fracture patients will have elevations due to the acute fracture. However, the investigators will attempt to obtain lab tests from the period prior to fracture to determine if they were normal. If unexplained elevations in alkaline phosphatase are found in labs prior to the fracture we will exclude that subject.
   7. Evidence of metastatic cancer or history of bone cancer or any active cancer other than basal or squamous cell carcinoma.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeri W Nieves, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data available for sharing 12-months after the publication of the primary paper. SAS datasets, a data dictionary, images of case report forms, SAS format library, the SAS program in which source data is recoded for analysis and data table summary descriptive statistics for data validation cross-check will be made available on an encrypted USB drive. A data sharing agreement is required.
Time Frame: 12 months after publication of results for 2 years
Access Criteria: Submission should be made to Nievesje@hss.edu

REFERENCES:
- [Result] Nieves JW, Cosman F, McMahon D, Redko M, Hentschel I, Bartolotta R, Loftus M, Kazam JJ, Rotman J, Lane J. Teriparatide and pelvic fracture healing: a phase 2 randomized controlled trial. Osteoporos Int. 2022 Jan;33(1):239-250. doi: 10.1007/s00198-021-06065-4. Epub 2021 Aug 12. PMID 34383100

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We included men and postmenopausal women >50 years of age within 1 month of acute pelvic fractures, occurring with minimal trauma. Sites included Hospital for Special Surgery, Helen Hayes Hospital or New York Presbyterian Hospital. Patients who had one or multiple pubic rami fractures (with or without sacral fractures) were included in the study. The first person was recruited into the study in May 2017 and the last person was recruited in August 2019.
Pre-assignment Details: Participants were excluded if they were unable to provide informed consent, if they were non-ambulatory prior to the fracture, or if they had a contraindication or intolerance to teriparatide. Serum calcium level had to be within normal range, serum creatinine could not be elevated more than 1.5 times above upper normal limit for age and alkaline phosphatase levels could not be greater than 1.5 times the upper normal limit.
Groups:
- Teriparatide: TPTD is supplied as a sterile, colorless, clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable delivery device (pen) for subcutaneous injection. Each prefilled delivery device is filled with 2.7 mL to deliver 2.4 mL. Each mL contains 250 mcg teriparatide (corrected for acetate, chloride, and water content), 0.41 mg glacial acetic acid, 0.1 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3 mg Metacresol, and Water for Injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4.
  Teriparatide Prefilled Syringe: TPTD 20 mcg
Period: 3 Month Endpoints- Blinded Portion
Arm/Group | Teriparatide | Placebo
Started | 18 | 17
Completed | 17 | 12
Not Completed | 1 | 5
Period: Open Label Extension 3 to 12 Months
Arm/Group | Teriparatide | Placebo
Started | 17 | 12
Completed | 12 | 9
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Participants must have taken at least one dose of study medication for intention to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Placebo | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.6 (8.1) | 81.0 (11.5) | 81.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 15 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (3.5) | 22.5 (5.5) | 22.3 (4.4)
history of fracture [Count of Participants; unit: Participants] | 12 | 12 | 24
multiple rami fractures [Count of Participants; unit: Participants] | 18 | 14 | 32
displaced fractures [Count of Participants; unit: Participants] | 8 | 9 | 17
sacral fractures [Count of Participants; unit: Participants] | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Evidence of Cortical Bridging for Fracture Healing
Description: Evidence of cortical bridging based on Focus CT,
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 18 | 15
Participants | 9 | 8

2. Secondary Outcome: Change in Pain by Numeric Rating Scale Between Baseline and Three Months
Description: Leads to a faster reduction in pain as assessed by the Numeric Rating Scale of 0 (no pain) to 10 (worst pain).
  The mean reduction in pain score from 0 to 3 months is reported. Higher scores mean a greater reduction in pain.
Time Frame: 3 months
Population: participants with a 3 month visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 17 | 12
score on a scale | 1.94 (3.42) | 2.78 (3.14)

3. Secondary Outcome: Functional Outcome Using a Battery That Includes Walking Speed, Repeated Chair Stands, and Balance at 3 Months
Description: More rapidly improved functional outcome using a short physical performance battery to assess lower extremity function (walking speed, repeated chair stands, and balance) at 3 months. Scale is 0 to 100 with higher scores indicating better physical performance.
Time Frame: 3 months
Population: All persons completing 3 month visit to provide data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 17 | 12
score on a scale | 74.2 (3.6) | 59.9 (4.7)

4. Secondary Outcome: Physical Function at 12 Months Using a Battery That Includes Walking Speed, Repeated Chair Stands, and Balance
Description: More rapidly improved functional outcome using a short physical performance battery to assess lower extremity function (walking speed, repeated chair stands, and balance) at 12 months. Scale is 0 to 100 with higher scores indicating better performance.
Time Frame: 12 months
Population: Participants providing 12 month data and taking study drug during extension
Measure: Mean (Standard Error); unit: score on a scale 0-100
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 10 | 7
score on a scale 0-100 | 70.0 (3.3) | 64.9 (4.1)

5. Secondary Outcome: Pain at 12 Months Based on the Numeric Rating Scale
Description: Pain at 12 months as assessed by the Numeric Rating Scale (0 to 10 where 0 means no pain and 10 worst pain)
Time Frame: 12 months
Population: Participants who completed 12 month visit
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 12 | 9
score on a scale | 1.5 (0.4) | 1.9 (0.6)

ADVERSE EVENTS:
Time Frame: One year
Groups:
- Teriparatide for 3 Months Then Open Label for 9 Months; Open Label Teriparatide Following Placebo: TPTD is supplied as a sterile, colorless, clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable delivery device (pen) for subcutaneous injection. Each prefilled delivery device is filled with 2.7 mL to deliver 2.4 mL. Each mL contains 250 mcg teriparatide (corrected for acetate, chloride, and water content), 0.41 mg glacial acetic acid, 0.1 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3 mg Metacresol, and Water for Injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4.
  Teriparatide Prefilled Syringe: TPTD 20 mcg
- Placebo for 3 Months: Placebo is supplied as a sterile, colorless, clear, isotonic solution in a glass cartridge which is pre-assembled into a disposable delivery device (pen) for subcutaneous injection. Each prefilled delivery device is filled with 2.7 mL to deliver 2.4 mL. Each mL contains 0.41 mg glacial acetic acid, 0.1 mg sodium acetate (anhydrous), 45.4 mg mannitol, 3 mg Metacresol, and Water for Injection. In addition, hydrochloric acid solution 10% and/or sodium hydroxide solution 10% may have been added to adjust the product to pH 4.
  Placebo: Matching placebo as a prefilled syringe with all inactive ingredients
Arm/Group | Teriparatide for 3 Months Then Open Label for 9 Months | Placebo for 3 Months | Open Label Teriparatide Following Placebo
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/18 | 1/17 | 3/12
Other Adverse Events (participants affected / at risk) | 12/18 | 4/17 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide for 3 Months Then Open Label for 9 Months (N=18) | Placebo for 3 Months (N=17) | Open Label Teriparatide Following Placebo (N=12)
cardiac (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
orthopedic procedure (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide for 3 Months Then Open Label for 9 Months (N=18) | Placebo for 3 Months (N=17) | Open Label Teriparatide Following Placebo (N=12)
Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
nausea vomiting diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
UTI (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
muscle or joint pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1) | 2 (2)
fatigue, loss of apatite, lethargy (Social circumstances) | 3 (3) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
bruising, blotching, squamous cell excision (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial had several limitations. The first is that we were underpowered to find an effect of TPTD on radiographic evidence of fracture healing due to a halt in supply of study medication, therefore, our findings should be considered exploratory. Recruitment was difficult; we screened 363 patients to recruit 35 subjects. It is also difficult to retain an older cohort with multiple underlying comorbidities. We only assessed healing at one time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02972424/Prot_SAP_000.pdf